CLINICAL TRIAL: NCT03751904
Title: Early Feasibility Study to Assess Safety and Device Performance of AcoustiCare™
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor is no longer pursuing the study.
Sponsor: Signature Medical, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SIG-0001
Record Dates: First submitted 2018-11-15; First posted 2018-11-23 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Heart Failure，Congestive
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AcoustiCare (Other): Single Arm
  Interventions: Device: AcoustiCare

INTERVENTIONS:
Device: AcoustiCare — Electronic stethoscope

SUMMARY:
AcoustiCareTM is a non-invasive clinical tool used for the detection of intracardiac pressures using heart sounds in patients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between the ages of 18 - 80 years
2. Willing and able to sign informed consent form
3. Normal subjects without a history of heart disease who are recruited from the surrounding community
4. Subjects with heart failure undergoing treatment in a hospital setting

Exclusion Criteria:

1. Hemodynamic instability (Systolic BP>180 or <90 and Diastolic BP>90 and <60)
2. Acute coronary syndrome
3. Prior heart transplant recipients
4. Subjects who are pacemaker dependent
5. Severe obesity (body mass index > 40 kg/m2)
6. Subjects who are pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2019-02-28 (Estimated); Study Completion 2019-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | Subjects will be assessed for adverse events through study completion, an average of 1 day
  The safety of the Acousticare device will be assessed by reviewing adverse events in all patients enrolled in the study